CLINICAL TRIAL: NCT01792245
Title: Topical Psoralen Ultraviolet Light A Versus Narrow Band Ultraviolet Light B Treatment for Recalcitrant Dermatoses of the Hand: A Prospective Randomized, Single-blinded Controlled Clinical Trial
Brief Title: Topical Psoralen Ultraviolet Light A Versus Narrow Band Ultraviolet Light B Treatment for Recalcitrant Dermatoses of the Hand
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: H12-02854
Record Dates: First submitted 2013-02-06; First posted 2013-02-15 (Estimated); Last update posted 2015-07-02 (Estimated); Status verified 2015-06

CONDITIONS: Vitiligo
Keywords: narrow band UVB; PUVA; psoriasis; eczema; hand
MeSH Terms: conditions — Vitiligo; Psoriasis; Eczema | interventions — Phototherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NB-UVB (Active Comparator): This single-blinded randomized bilateral left to right controlled comparison clinical trial of 24 weeks duration will compare the efficacy of NB-UVB to t-PUVA. For each patient one hand will be randomly assigned to receive t-PUVA and the other hand will receive NB-UVB. Each hand will receive treatment with either NB-UVB or topical PUVA three times weekly. Treatment will be performed until complete or almost complete clearing of psoriasis/eczema or until 50 exposures (over 16 weeks) have been reached, whichever comes first.
  Interventions: Device: Phototherapy
- Topical PUVA (Active Comparator): This single-blinded randomized bilateral left to right controlled comparison clinical trial of 24 weeks duration will compare the efficacy of NB-UVB to t-PUVA. For each patient one hand will be randomly assigned to receive t-PUVA and the other hand will receive NB-UVB. Each hand will receive treatment with either NB-UVB or topical PUVA three times weekly. Treatment will be performed until complete or almost complete clearing of psoriasis/eczema or until 50 exposures (over 16 weeks) have been reached, whichever comes first.
  Interventions: Device: Phototherapy

INTERVENTIONS:
Device: Phototherapy

SUMMARY:
Hand psoriasis/eczema is a common problem which is characterized by itchy, erythematous and scaly lesions often with a long lasting and relapsing course. Treatment is difficult with considerable number of patients do not or only partially respond to the current treatments. Several studies have shown the therapeutic effectiveness of the combination of topical psoralen with long wavelength ultraviolet A radiation (PUVA) in treating hand psoriasis/eczema. Topical PUVA is has several short- and long-term side effects. Narrow band ultraviolet B (NB-UVB) has emerged recently as an important treatment for a variety of photoresponsive diseases including psoriasis and eczema. For most conditions (other than hand psoriasis/eczema) NB-UVB has been shown to have similar therapeutic results to PUVA with less side effects. There are only a few studies published on the efficacy of NB-UVB for hand psoriasis/eczema. Therefore, this study is aimed at comparing the efficacy and safety of t-PUVA and NB-UVB in treating these conditions.

DETAILED DESCRIPTION:
Hand dermatoses is a common problem which is characterized by itchy, erythematous and scaly lesions often with a long lasting and relapsing course. Patients presenting with these severe cutaneous changes are classified as having severe recalcitrant hand dermatoses. Treatment is difficult with considerable number of patients do not or only partially respond to the current treatments. Current treatment regimens mainly involve the use of high potency topical corticosteroids, which has only limited affect. Systemic treatment modalities have been utilized but have serious side effects with limited improvement of disease.

Several studies have shown the therapeutic effectiveness of the combination of topical psoralen with long wavelength ultraviolet A radiation (PUVA) in treating hand dermatoses. Topical PUVA is commonly associated with mild local sunburn reactions that often necessitate temporarily withholding treatment or decreasing the light dose. This subsequently leads to a delay in response or a prolongation of the treatment. Long term side effects include aging of the skin, hyperpigmentation, and a small increased risk of skin cancer that is more common in systemic PUVA. Narrow band ultraviolet B (NB-UVB) has emerged recently as an important treatment for a variety of photoresponsive diseases including psoriasis and eczema. For most conditions (other than hand psoriasis/eczema) NB-UVB has been shown to have similar therapeutic results to PUVA with less side effects.

There are only a few studies published on the efficacy of NB-UVB for hand psoriasis/eczema. Our hypothesis is that NB-UVB and topical PUVA will result in at least comparable improvement in hand psoriasis/eczema with less side effects associated with NB-UVB. We plan on conducting a prospective single-blind randomized clinical trial to compare the efficacy and safety of topical PUVA and NB-UVB in treating hand psoriasis/eczema.

Study Objectives

1. To compare the effect of topical PUVA and NB-UVB on visual cutaneous symptoms in patients presenting with recalcitrant hand dermatoses.
2. To compare the side effect profile of topical PUVA and NB-UVB when treating patients with recalcitrant hand dermatoses.

ELIGIBILITY:
Inclusion Criteria:

* Chronic symmetrical severe hand psoriasis and eczema (allowing up to 15% difference in surface area between both hands). These include patients that have received topical corticosteroids previously and may or may have not responded to treatment.
* Subjects should be 18 years old or older.

Exclusion Criteria:

* Any serious medical illness that will restrict the patient's ability to receive light treatments. That includes skin conditions, such as skin cancer or severe blistering conditions, or any serious medical conditions affecting the sensation of the extremities (eg. diabetic neuropathy, cervical stenosis).
* Patients known to have a photosensitivity disorder
* Patients with a history of intolerance to UVB and/or UVA light therapy.
* Any subject who is on treatment or was on treatment for hand psoriasis/eczema less than two (topical) or four (systemic/phototherapy) weeks prior to enrollment in the study.
* Pregnancy or breast-feeding.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2013-02; Primary Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
The primary endpoint will be based on the change in visual cutaneous symptoms as measured by the modified ASI score | Baseline, every four weeks up to 16 weeks, and at 24 weeks

SECONDARY OUTCOMES:
The overall change in physical appearance of the hand will be assessed by the global assessment | Every four weeks up to 16 weeks, and at 24 weeks
Adverse effects will be assessed every four weeks, including erythema, pruritus, and tanning. This will be assessed using the following scale: 0=none, 1=mild, 2=moderate, 3=severe. | Every four weeks up to 16 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Harvey Lui, MD, FRCPC, Principal Investigator — University of British Columbia
Locations (1):
- The Skin Care Center, Vancouver General Hospital, Vancouver, British Columbia, Canada